CLINICAL TRIAL: NCT06665152
Title: Comparison of Postoperative Pain After Root Canal Preparation With Reciprocal (WaveOne) Versus Continuous Rotary (ProTaper Gold) For Asymptomatic Irreversible Pulpitis
Brief Title: Comparison of Post-operative Pain After Using Different File Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Abdullah (Other)
Responsible Party: Sponsor-Investigator, Ahmed Abdullah, Principal investigator, Armed Forces Institute of Dentistry, Pakistan
Organization: Armed Forces Institute of Dentistry, Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMHLMCIOD
Record Dates: First submitted 2024-10-26; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Comparison of postoperative pain in two groups of patients, who underwent root canal treatment with two different file systems. total 74 patients divided into two groups and given different interventional treatment to monitor pain after treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients did not know which file system was used in their treatment. The investigator was also not disclosed the intervention's name; rather, a code name was given to them.
  Outcomes accessor also did not know the exact name but was provided with a code name.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ProTaper Group (Experimental): These patients underwent root canal treatment due to pain in their molar teeth. The file system used in this arm was ProTaper (Dentsply), a rotary file system that moves in a complete 360° rotation and prepares a root canal.
  Interventions: Device: ProTaper File System
- WaveOne Group (Active Comparator): These patients underwent root canal treatment due to pain in their molar teeth. The file system used in this arm was WaveOne(Dentsply), a reciprocating file system that moves in 150° anticlockwise and 30° clockwise motion and prepares a root canal.
  Interventions: Device: WaveOne File System

INTERVENTIONS:
Device: ProTaper File System — A rotary file system
  Arms: ProTaper Group
Device: WaveOne File System — A reciprocating file system
  Arms: WaveOne Group

SUMMARY:
To compare the postoperative pain in patients undergoing root canal instrumentation with two different file systems, WaveOne and ProTaper systems.

DETAILED DESCRIPTION:
Endodontic postoperative pain is experienced after the procedure of root canal. It is defined as an unpleasant sensation, of varying degree, experienced by the patients. Depending upon the individual and other variable, the range of postoperative pain lies between 3% to 58%. Endodontic postoperative pain could occur due to various factors that can be microbial, injured pulp, chemical, or mechanical. Factors that influence pain following a root canal include the presence of preoperative pain, apical debris extrusion, intracanal interappointment dressing extrusion, presence of periapical pathosis, hyper occlusion, and irrigant extrusion.

Although apically extruded debris can be reduced through various means, it cannot be completely avoided. Thus, increasing the incidence of postoperative pain in patients. The debris produced during apical extrusion contains necrotic tissue, dental chips, microbes, pulp tissue, and canal irrigants. The infected debris may disturb the balance between the microbes and the immune system, leading to acute exacerbation.

Manual steel K files tend to produce more debris, causing a high risk of postoperative discomfort. Nickel-titanium rotary instruments powered by the engine have various advantages including; time-saving, preservation of root canal anatomy, and homogeneous preparation of the shape of the root canal. The debris produced by these instruments is potentially lesser than the manual files. Mainly because they have rotary action and they excavate the debris with the help of their flutes. Repeated irrigation along with the action of an engine-driven instrument, has the potential to decrease postoperative pain. WaveOne reciprocating file instruments have potential advantages including reduced fatigue, resistance to fracture, less debris extrusion, good shaping ability, no cross-contamination (single use), and reduced cost.

Relation between debris extrusion and postoperative care has not been established in any previous study. This study is aimed at comparing the use of ProTaper Universal and WaveOne system, for preparation of permanent human teeth during root canal procedure and their effect on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unremarkable/ noncontributory medical history
2. Healthy persons between the ages of 18 and 60 years
3. Maxillary and mandibular molar teeth diagnosed with symptomatic irreversible pulpitis.
4. Patients not having taken any medication for 6 hours before treatment
5. No allergies to the drugs or dental material being used in the treatment

Exclusion Criteria:

1. Patients who had taken analgesics on anti-inflammatory drugs within the last 12 hours
2. Pregnant women and patients with immunocompromised health state
3. Patients having severe malocclusion associated with traumatic occlusion
4. Teeth with calcified canals
5. Teeth with periapical radiolucency
6. Teeth with root resorption
7. Teeth previously undergone root canal treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 6 hours - 72 hours
  Document and compare post-operative pain after root canal treatment, after using two different motorized file systems with different mechanisms. The Visual Analog scale (VAS) would be used to assess the pain. The patients would be guided in detail about the VAS scoring system and mark pain according to the readings on VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem A Rana, BDS, FCPS, Study Director — CMH LMC IOD
Locations (1):
- 28 MDC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
individual participant data to not be disclosed due to privacy reasons and data sharing for statistical analysis to be done with codenames.